CLINICAL TRIAL: NCT00909077
Title: A Randomised Phase III Study of the Efficacy of High Dose Dexamethasone Versus High Dose Dexamethasone in Combination With Rituximab (MabThera®)in Patients With Newly Diagnosed Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: The Efficacy of Dexamethasone Versus Dexamethasone Combined With Rituximab in Patients With Newly Diagnosed Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Forskningsenheden, Forskningsenhed, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Rituximab-DXM
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP-Rituximab-dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Combination therapy with Dexamethasone and Rituximab
  Interventions: Drug: Dexamethasone and Rituximab
- 2 (Active Comparator): Dexamethasone as monotherapy
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone tablets: 40 mg/day for four days
  Arms: 2
Drug: Dexamethasone and Rituximab — Dexamethasone tablets: 40 mgs/day for four days Rituximab iv 375 mg/m^2 weekly, a total of four times. Administered on day 2 (i.e. the patient has been treated with Dexamethasone for one day)
  Arms: 1

SUMMARY:
In this study we want to investigate if combination therapy with rituximab (R) + dexamethasone (DXM) is superior to monotherapy with DXM in patients with newly diagnosed idiopathic thrombocytopenic purpura (ITP). Before treatment molecular studies - gene expression profiling - are performed to characterize at the molecular level those patients responding adequately to the treatment as compared to those obtaining a minor or no responses.

The hypothesis is that combination therapy is superior to monotherapy as defined above. Using gene expression studies up-front the hypothesis is that this method may be able to predict the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Diagnosis = ITP + platelet count above or equal to 25 Mia/l or platelet count above or equal to 50 Mia/l and bleeding from the mucous membranes.
* Adequate contraceptive measures within the last 3 months for women of childbearing potential.

Exclusion Criteria:

* Performance status above or equal to 2
* Previous treatment with rituximab
* Immunosuppressive treatment within the last month except for not previously treated patients
* Other serious disease
* Pregnant women and nursing mothers
* Contraindication for rituximab treatment.
* Active infection requiring antibiotic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2004-08 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained partial response after 6 months | 6 months

SECONDARY OUTCOMES:
Remission rates in the 2 arms at day 7, 10, 14,21, 28, month 2 - 12, year 2 - 5 | day 7, 10, 14,21, 28, month 2 - 12, year 2 - 5

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Hasselbalch, MD, Principal Investigator — Copenhagen University Hospital Herlev, Department of Haematology
Locations (10):
- Denmark (10):
  - Aalborg Hospital, Aalborg
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Copenhagen University Hospital Herlev, Department of Haematology, Herlev
  - Regional Hospital Holstebro, Holstebro
  - Naestved Hospital, Næstved
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Vejle Hospital, Vejle
  - Viborg Hospital, Viborg

REFERENCES:
- [Derived] Gudbrandsdottir S, Birgens HS, Frederiksen H, Jensen BA, Jensen MK, Kjeldsen L, Klausen TW, Larsen H, Mourits-Andersen HT, Nielsen CH, Nielsen OJ, Plesner T, Pulczynski S, Rasmussen IH, Ronnov-Jessen D, Hasselbalch HC. Rituximab and dexamethasone vs dexamethasone monotherapy in newly diagnosed patients with primary immune thrombocytopenia. Blood. 2013 Mar 14;121(11):1976-81. doi: 10.1182/blood-2012-09-455691. Epub 2013 Jan 4. PMID 23293082